CLINICAL TRIAL: NCT04219228
Title: A Prospective School-based Study of Myopia in Children in Southern China
Brief Title: Zhaoqing Myopia Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Other Study IDs: 2019KYPJ171
Record Dates: First submitted 2019-12-28; First posted 2020-01-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Wearable Electronic Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Students in urban counties: All first-grade students in urban counties will undergo anthropometry and ophthalmic examination, and be required to complete questionnaires and wear wearable devices to collect environmental information and daily activities.
  Interventions: Diagnostic Test: Ophthalmic examinations; Device: Wearable devices
- Students in rural counties: All first-grade students in rural counties will undergo anthropometry and ophthalmic examination, and be required to complete questionnaires and wear wearable devices to collect environmental information and daily activities.
  Interventions: Diagnostic Test: Ophthalmic examinations; Device: Wearable devices

INTERVENTIONS:
Diagnostic Test: Ophthalmic examinations — Ophthalmic examinations include visual acuity, cover test and ocular dominance, noncycloplegic autorefraction, cycloplegia, ocular biometric measurements, cycloplegic auto-refraction, subjective refraction, and anterior and posterior segment examination.
Device: Wearable devices — Physical activity, light intensity, and visual information will be measured with wearable devices.

SUMMARY:
Myopia is a common cause of vision loss, being particularly prevalent in children in East and Southeast Asia. The investigators will assess prevalence and incidence of myopia, identify digital biomarkers associated with myopia, and validate algorithms for the detection and/or predition of myopia and other ocular abnormalities in school-aged children in both urban and rural settings in Southern China.

DETAILED DESCRIPTION:
Myopia is a common cause of vision loss, being particularly prevalent in East and Southeast Asia. It is still not entirely clear whether and how visual experience in an urban environment with less outdoor exposure could have an impact on the development and progression of myopia. Zhaoqing has a relatively stable population of 4,084,600, which are representative of the Chinese population in term of demographic and socioeconomic characteristics.

Therefore, the investigators will conduct a longitudinal cohort study in both urban and rural settings to examine prevalence and incidence of myopia, identify digital biomarkers associated with myopia, and validate algorithms for the detection and/or predition of incidence and progression of myopia and other ocular abnormalities in school-aged children in Zhaoqing.

ELIGIBILITY:
Inclusion Criteria:

* All first-grade students from 10 primary schools in urban counties, and from 10 primary schools in rural counties, Zhaoqing city.

Exclusion Criteria:

* No.

Ages: 6 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: All first-grade students from 10 primary schools in urban counties, and from 10 primary schools in rural counties, Zhaoqing city.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2019-12-14 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-02-02 (Estimated)

PRIMARY OUTCOMES:
Incident myopia | 3 years
  Incident myopia is defined as myopia detected during follow up among those without myopia at baseline. Myopia is defined as any eye's SER (sphere + 1/2 cylinder) of at least -0.5 diopters (D).

SECONDARY OUTCOMES:
Prevalence of myopia | baseline
  Myopia is defined as any eye's SER (sphere + 1/2 cylinder) of at least -0.5 diopters (D).
Change in axial length | 1 year, 2 years, 3 years
  Axial length will be measured with a non-contact optical device.
Prevalence of amblyopia, strabismus and other ocular abnormalities | baseline
  Cover-uncover tests will be performed to detect strabismus. Any ocular abnormalities, including corneal opacities, lens opacities, and retinal diseases will be recorded based on slit lamp, direct ophthalmoscopic and/or mobile phone video examination. Participants with an uncorrected visual acuity 6/7.5 or worse with undergo subjective refraction to identify amblyopia.
Area under the receiver operating characteristic curve of the deep learning algorithm for the prediction of incident myopia | 1 year
  The investigators will estimate the area under the receiver operating characteristic curve of the deep learning algorithm for the prediction of incident myopia.
Sensitivity and specificity of the deep learning algorithm for the prediction of incident myopia | 1 year
  The investigators will estimate sensitivity and specificity of the deep learning algorithm for the prediction of incident myopia.
Area under the receiver operating characteristic curve of the deep learning algorithm for the prediction of fast progressing myope | 1 year
  The investigators will estimate the area under the receiver operating characteristic curve of the deep learning algorithm for the prediction of fast progressing myope (a change in SER of 0.75D or more per year).
Sensitivity and specificity of the deep learning algorithm for the prediction of fast progressing myope | 1 year
  The investigators will estimate the sensitivity and specificity of the deep learning algorithm for the prediction of fast progressing myope (a change in SER of 0.75D or more per year). Cycloplegic spherical refraction changes measured by an auto-refractometer will be used as the indicator of myopia progression.
Area under the receiver operating characteristic curve of the diagnostic algorithm in identifying abnormal vision screening result | baseline
  The investigators will estimate the area under the receiver operating characteristic curve of the diagnostic algorithm in identifying abnormal vision screening result (e.g., abnormal eye lid, abnormal cornea, and strabismus detected with mobile devices).
Sensitivity and specificity of the diagnostic algorithm in identifying abnormal vision screening result | baseline
  The investigators will estimate the sensitivity and specificity of the diagnostic algorithm in identifying abnormal vision screening result (e.g., abnormal eye lid, abnormal cornea, and strabismus detected with mobile devices).
Post-vision screening referral uptake | 3 months
  Any referral uptake will be confirmed by telephone follow-up.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong
  - Schools, Zhaoqing, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morgan IG, Ohno-Matsui K, Saw SM. Myopia. Lancet. 2012 May 5;379(9827):1739-48. doi: 10.1016/S0140-6736(12)60272-4. PMID 22559900
- [Result] Zadnik K, Mutti DO. Outdoor Activity Protects Against Childhood Myopia-Let the Sun Shine In. JAMA Pediatr. 2019 May 1;173(5):415-416. doi: 10.1001/jamapediatrics.2019.0278. No abstract available. PMID 30907935
- [Result] Ojaimi E, Rose KA, Smith W, Morgan IG, Martin FJ, Mitchell P. Methods for a population-based study of myopia and other eye conditions in school children: the Sydney Myopia Study. Ophthalmic Epidemiol. 2005 Feb;12(1):59-69. doi: 10.1080/09286580490921296. PMID 15848921
- [Result] Li SM, Liu LR, Li SY, Ji YZ, Fu J, Wang Y, Li H, Zhu BD, Yang Z, Li L, Chen W, Kang MT, Zhang FJ, Zhan SY, Wang NL, Mitchell P; Anyang Childhood Eye Study Group. Design, methodology and baseline data of a school-based cohort study in Central China: the Anyang Childhood Eye Study. Ophthalmic Epidemiol. 2013 Dec;20(6):348-59. doi: 10.3109/09286586.2013.842596. Epub 2013 Oct 25. PMID 24160405
- [Result] He M, Zheng Y, Xiang F. Prevalence of myopia in urban and rural children in mainland China. Optom Vis Sci. 2009 Jan;86(1):40-4. doi: 10.1097/OPX.0b013e3181940719. PMID 19104465
- [Result] Negrel AD, Maul E, Pokharel GP, Zhao J, Ellwein LB. Refractive Error Study in Children: sampling and measurement methods for a multi-country survey. Am J Ophthalmol. 2000 Apr;129(4):421-6. doi: 10.1016/s0002-9394(99)00455-9. PMID 10764848
- [Derived] Chen X, Ye G, Zhong Y, Jin L, Liang X, Zeng Y, Zheng Y, Lan M, Liu Y. Prevalence, incidence, and risk factors for myopia among urban and rural children in southern China: protocol for a school-based cohort study. BMJ Open. 2021 Nov 5;11(11):e049846. doi: 10.1136/bmjopen-2021-049846. PMID 34740929